CLINICAL TRIAL: NCT02066233
Title: Prospective Study to Compare the Efficacy of E.G.Scan to Detect Barrett's Esophagus Compared With Standard Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: IntroMedic Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Prasad G. Iyer, Associate Professor of Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-008214
Record Dates: First submitted 2014-02-03; First posted 2014-02-19 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's; esophagus; reflux; heartburn; screening
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Subjects with Barrett's Esophagus (Active Comparator): All subjects will receive transnasal endoscopy (EG Scan II) followed by standard endoscopy.
  Interventions: Device: EG Scan II (transnasal endoscopy); Procedure: Standard Endoscopy
- Subjects with Reflux and/or Heartburn (Active Comparator): All subjects will receive EG Scan II (transnasal endoscopy) followed by standard endoscopy.
  Interventions: Device: EG Scan II (transnasal endoscopy); Procedure: Standard Endoscopy

INTERVENTIONS:
Device: EG Scan II (transnasal endoscopy)
Procedure: Standard Endoscopy

SUMMARY:
The purpose of this study was to evaluate whether a disposable nasal endoscope called "E.G. Scan II" will visualize the esophagus as well as the standard test, sedated endoscopy.

DETAILED DESCRIPTION:
All subjects underwent two procedures: the E.G.Scan II followed by standard endoscopy in a tandem design. The E.G. Scan II is a transnasal endoscope system to capture and transmit images of the esophagus. Captured images can be reviewed via the E.G. View for diagnosis of diseases related to the esophagus. Generally, the commercial esophagoscope system has reusable probes, but E.G. Scan™ II has a single use probe because reusable probes have the risk of infection and pollution.

Prior to the E.G.Scan, subjects received a standard prep for the procedure. The two procedures were performed by two different experienced endoscopists who were blinded to the indication of the procedure. At both procedures a note was made of any abnormality of the esophagus. Every subject with an endoscopic diagnosis of Barrett's Esophagus had clinical biopsies taken to confirm diagnosis. Subject tolerability was measured with a 10-point visual analog scale (VAS) where 0 represented the "worst experience" and 10 the "best experience."

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants aged 18 years or above who are scheduled for routine upper GI endoscopy for Barrett's Esophagus surveillance, varices surveillance and dyspepsia.
2. Able and willing to give informed consent.

Exclusion Criteria:

1. Patients known to be intolerant to endoscopy.
2. Patients with frequent epistaxis.
3. Patients not clinically fit for endoscopy as judged by their care team.
4. Pregnant women.
5. Patients with allergy/sensitivity to Simethicone (Mylicon), Phenylephrine, Lidocaine nasal spray, Benzocaine spray (Topex)
6. Use of anticoagulants or antiplatelets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prasad G Iyer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sami SS, Iyer PG, Pophali P, Halland M, di Pietro M, Ortiz-Fernandez-Sordo J, White JR, Johnson M, Guha IN, Fitzgerald RC, Ragunath K. Acceptability, Accuracy, and Safety of Disposable Transnasal Capsule Endoscopy for Barrett's Esophagus Screening. Clin Gastroenterol Hepatol. 2019 Mar;17(4):638-646.e1. doi: 10.1016/j.cgh.2018.07.019. Epub 2018 Aug 3. PMID 30081223

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Barrett's Esophagus; Subjects With Reflux and/or Heartburn: All subjects will receive EG Scan II (transnasal endoscopy) followed by standard endoscopy.
Period: EG Scan II (Day 1)
Arm/Group | Subjects With Barrett's Esophagus | Subjects With Reflux and/or Heartburn
Started | 50 | 50
Completed | 44 | 44
Not Completed | 6 | 6
Not completed — difficulty intubating subject | 6 | 6
Period: Standard Endoscopy (Day 2)
Arm/Group | Subjects With Barrett's Esophagus | Subjects With Reflux and/or Heartburn
Started | 44 | 44
Completed | 44 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects With Barrett's Esophagus | Subjects With Reflux and/or Heartburn | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.66 (11.62) | 51.72 (15.07) | 56.19 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 20 | 29
  Male | 41 | 30 | 71
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Median Tolerability Score on 10-point Visual Analog Scale (VAS)
Description: On the 10-point VAS, 0 represented the "worst experience" and 10 the "best experience."
Time Frame: Within 48 hours
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Subjects With Barrett's Esophagus | Subjects With Reflux and/or Heartburn
Number analyzed (Participants) | 44 | 44
units on a scale
  EG II Scan | 7 [3 to 10] | 8 [1 to 10]
  Standard Endoscopy | 8 [4 to 10] | 8 [2 to 10]

2. Secondary Outcome: Preference for Either of the Two Procedures, EG II Scan Versus Standard Endoscopy
Description: Subjects were asked the following question: "Based on the overall experience (including need for sedation, ability to drive, time off work, procedure comfort, procedure time, etc.). Which procedure would you prefer to have in the future?" Possible answers were: Nasal camera test (EG), oral camera test (Gastroscopy), or either test.
Time Frame: Two weeks
Population: Two subjects on the reflux and/or heartburn arm didn't answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Barrett's Esophagus | Subjects With Reflux and/or Heartburn
Number analyzed (Participants) | 42 | 44
Participants
  Nasal Camera Test | 21 | 18
  Oral Camera Test | 4 | 11
  Either Test | 17 | 15

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Presenting adverse events per per intervention was not possible, as most patients were sedated prior to the procedures and only a few were not sedated. Therefore the adverse events were per patient population (study arm).
Arm/Group | Subjects With Barrett's Esophagus | Subjects With Reflux and/or Heartburn
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 44/44 | 44/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Barrett's Esophagus (N=44) | Subjects With Reflux and/or Heartburn (N=44)
Gagging/Retching (Gastrointestinal disorders) | 32 (32) | 36 (36)
Choking (Gastrointestinal disorders) | 21 (21) | 12 (12)
Discomfort (General disorders) | 38 (38) | 43 (43)
Nasal Pain (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 34 (34)
Nose Bleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes